CLINICAL TRIAL: NCT00474097
Title: Follow-Up Phone Calls After Colorectal Surgery to Assess Patient Satisfaction and Post-Operative Outcomes
Brief Title: Follow-Up Phone Calls After Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Conor Delaney, MD, PhD, Principal Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: 01-06-03
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Colorectal Surgery; Colorectal Neoplasms; Colitis, Ulcerative; Diverticulitis; Colonic Polyps
Keywords: Colorectal Neoplasms; Colitis, Ulcerative; Diverticulitis; Colonic Polyps; Crohn Disease
MeSH Terms: conditions — Colorectal Neoplasms; Colitis, Ulcerative; Diverticulitis; Colonic Polyps; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess if follow-up telephone calls after colorectal surgery affects a patient's satisfaction, the outcome of their surgery, and their quality of life. In addition, readmissions, complications and emergency room visits can be tracked via these telephone calls, ensuring optimal communication between patients and the surgical office.

DETAILED DESCRIPTION:
Follow-up with patients after surgery is necessary to assess levels of rehabilitation, answer questions and expresses an attitude of caring, as well as assist in marketing procedures for the hospital or institution (Fallis, 2001). Surveillance after discharge from the hospital may be difficult as most patients are no longer monitored by health care professionals. If home health care is not required, the patient may not have contact with his/her doctor or nurse until the follow-up appointment which frequently is 4- 6 weeks post surgery.

There is evidence in the literature that telephone contact is beneficial for patients. The strongest and most current evidence came from a meta-analysis by Meade (2004) on research supporting phone calls post-operatively for hospitalized patients. This analysis provided a significant and valid review of health care professionals providing this service, looking at various patient populations and different hospital settings. 29 articles were published from 1981 to 2004 and reviewed to gather a compilation of research findings in this area. Regardless of the design of the research, the findings suggest that follow-up phone calls to patients after discharge provide invaluable opportunities to enhance practice in the following areas: Appraisal and evaluation of patient education, Practice improvement trends, Quality of care, Medication compliance and adherence to discharge instructions, Evaluation of overall hospital performance.

There is no evidence specifically addressing telephone contact after discharge in the colorectal surgery population which will be the basis of this study. Nurses providing follow-up phone calls to patients in the early post operative phase may assist in preventing or minimizing the effects of postoperative complications by reinforcing discharge instructions, answering patients' questions, and assessing their concerns. Potential serious complications may therefore be addressed early.

The purpose of this study is to assess if follow-up telephone calls after surgery affects patient satisfaction, surgical outcomes and quality of life in the early post-operative phase after colorectal surgery. In addition, tracking of readmissions, complications and emergency room visits via telephone calls can ensure communication between the patients and the surgical office is optimal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years of age and older
* Subjects of either sex
* Subjects who will undergo any moderate or major colorectal surgery requiring an overnight hospital stay at University Hospitals Case Medical Center
* Subjects who agree to participate in the study program and provide written informed consent
* Diagnoses such as Crohn's disease, ulcerative colitis, rectal or colon cancer, colon or rectal polyps and diverticulitis

Exclusion Criteria:

* Patients in the middle of three part surgery or had recent surgery (i.e., back for stoma closure for J-pouch)
* Patients with diagnosis of rectal prolapse, condyloma, and any conditions that require non-invasive outpatient procedures
* Pregnant women, minors, psychiatric patients and prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal Surgery clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
to assess if follow-up telephone calls after surgery affects patient satisfaction, surgical outcomes and quality of life in the early post-operative phase after colorectal surgery | not specific

SECONDARY OUTCOMES:
to track readmissions, complications and emergency room visits via telephone calls to ensure communication between the patients and the surgical office is optimal. | not specific

CONTACTS AND LOCATIONS:
Overall Officials: Conor Delaney, MD, PhD, Principal Investigator — University Hospitals of Cleveland/ Institute for Surgical Innovation
Locations (1):
- University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio, United States